CLINICAL TRIAL: NCT01140256
Title: Longitudinal Zinc Intakes and Exchangeable Zinc Pool Sizes in Breastfed Small for Gestational Age vs Appropriate for Gestational Age Infants in Pakistan
Acronym: EZP
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Collaborators: International Atomic Energy Agency (Other Government); University of Colorado, Denver (Other)
Responsible Party: Shabina Ariff, Aga Khan University
Other Study IDs: 585-Ped/ERC-06
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2009-07

CONDITIONS: Micronutrients; Gestational Age
Keywords: Zinc; SGA; AGA; stable isotope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- SGA infants: SGA infants were recruited at birth and zinc stable isotope was administered at birth and at 6 months of age .This was a longitudinal study whereby the growth trajectory and zinc pools were measured.
- AGA: AGA infants were recruited at birth and zinc stable isotope was administered at birth and at 6 months of age .This was a longitudinal study whereby the growth trajectory and zinc pools were measured.
- SGA infant: Infants who were born small for gestational age were recruited and zinc stable isotopes were administered at birth and at 6 months.

SUMMARY:
Large-scale zinc supplementation studies have demonstrated highly significant positive effects on growth, morbidity and mortality in infants who are born small for gestational age (SGA). This suggests these infants may have higher postnatal requirements compared to appropriate for gestational age (AGA) infants, possibly due to inadequate zinc intake from breast milk due either to lower volume or to differences in milk zinc concentrations from mothers of SGA compared to AGA infants. Alternatively, SGA infants may have lower zinc stores at birth, which may reflect a greater postnatal requirement for optimal zinc status. It is thus possible that the zinc requirements of the SGA infant exceed the zinc intake that can be achieved from exclusive breastfeeding, which is recommended for the first 6 mo of life. The exchangeable zinc pool (EZP) is defined as the estimate of the total size of the combined pools of zinc that exchange with zinc in plasma within approximately 2-3 days and may also differ between SGA and AGA infants.

1. Compare longitudinal zinc intake by measuring milk zinc concentrations and volume of intake of breast milk between SGA and AGA infants through first 12 mo.
2. Compare post-natal growth rates for SGA and AGA infants through the first 12 mo of life in relation to zinc intake.
3. Compare size of exchangeable zinc pool (EZP) at birth and at 6 mo of age between SGA and AGA infants.

Hypotheses:

1. Zinc concentrations in human milk will not be significantly different at any stage of lactation between mothers of SGA infants and mothers of AGA infants.
2. The volume of breast milk intake relative to body weight will be similar between SGA and AGA infants, but the total intake will be lower in SGA infants.
3. Linear growth rates, rate of weight gain, and rate of growth in head circumference will be significantly lower in infants born SGA, and will be positively correlated with total daily zinc intake.
4. The size of the EZP at birth will be significantly smaller in absolute size and relative to body weight in infants born SGA compared to AGA

DETAILED DESCRIPTION:
Scientific Background:

Large-scale zinc supplementation studies have demonstrated highly significant positive effects on growth, morbidity and mortality in infants who are born small for gestational age (SGA). This suggests these infants may have higher postnatal requirements compared to appropriate for gestational age (AGA) infants, possibly due to inadequate zinc intake from breast milk due either to lower volume or to differences in milk zinc concentrations from mothers of SGA compared to AGA infants. Alternatively, SGA infants may have lower zinc stores at birth, which may reflect a greater postnatal requirement for optimal zinc status. It is thus possible that the zinc requirements of the SGA infant exceed the zinc intake that can be achieved from exclusive breastfeeding, which is recommended for the first 6 mo of life. Estimated rates of infants born with intrauterine growth retardation, including SGA, are 25-40% of all births in south Asia (Bhutta - 2004a).

Scientific Scope of the Project (Scientific problems to be addressed with overall and specific objectives):

The overall objective of this project is to compare zinc intake from human milk and other fluids and complementary foods in SGA and AGA infants through the first 12 mo of life; growth for each group will also be monitored. A secondary goal is to compare the size of the exchangeable zinc pool in SGA and AGA infants at birth and at 6 mo, the period of recommended exclusive breastfeeding.

Specific Aims:

1. Compare longitudinal zinc intake by measuring milk zinc concentrations and volume of intake of breast milk between SGA and AGA infants through first 12 mo.
2. Compare post-natal growth rates for SGA and AGA infants through the first 12 mo of life in relation to zinc intake.
3. Compare size of exchangeable zinc pool (EZP) at birth and at 6 mo of age between SGA and AGA infants.

Expected Outcomes:

Expected outcomes include longitudinal data from SGA and AGA infants during the first year of life, including human milk intake, zinc concentrations in human milk, zinc intake from human milk, estimated intake of non-milk fluids and complementary foods, anthropometric measurements (length, weight, and head circumference), and size of exchangeable zinc pool; cross-sectional data on plasma zinc, ferritin and hemoglobin at 6 mo will also be obtained. These outcomes will all be compared between SGA and AGA infants. Relationships among variables will also be examined, including relationship of zinc intake and size of EZP to observed growth outcomes.

ELIGIBILITY:
Inclusion Criteria:

Mothers: Healthy women 18-40 yr; primips or multips; Infants: Healthy at birth

Exclusion Criteria:

Mothers: tobacco or alcohol use during pregnancy; HIV or chronic infection such as TB.

Infants: twins/multiples; congenital infections, malformations; gestational age < 37 wk ; severe anemia at birth.

-

Max Age: 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: SGA and AGA infants born to healthy mothers.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-01; Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To Compare size of exchangeable zinc pool (EZP) at birth and at 6 mo of age between SGA and AGA infants
  We measured the exchangeable zinc pool sizes in exclusively breast fed infants at birth and then at 6 months of age among the SGA and AGA infants by zinc stable isotope technique.Intravenous dose of pre measured was administered.Urine was collected and analyzed for enrichemnt of zinc isotope.The entire procedure was repeated at 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan university, Karachi, Sindh, Pakistan